CLINICAL TRIAL: NCT02560779
Title: An Open Label Phase 1B/2 Trial of TRC105 and Sorafenib in Patients With Hepatocellular Carcinoma (HCC)
Brief Title: Trial of TRC105 and Sorafenib in Patients With HCC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105HCC101
Record Dates: First submitted 2015-09-10; First posted 2015-09-25 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: TRC105; CD105; Endoglin; Angiogenesis inhibitor; HCC; TKI; Tyrosine Kinase Inhibitor; Sorafenib; Nexavar
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — carotuximab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carotuximab (TRC105) and Sorafenib (Experimental): Carotuximab (TRC105) in combination with standard dose Sorafenib.
  Interventions: Drug: Carotuximab (TRC105); Drug: Sorafenib

INTERVENTIONS:
Drug: Carotuximab (TRC105) — Bi-weekly iv TRC105 (15 mg/kg) will be given with 400mg sorafenib twice daily in the phase 1B portion of the study. Weekly iv TRC105 (10 mg/kg) will be given with 400mg sorafenib twice daily in the phase 2 portion of the study.
  Other Names: Chimeric Antibody (TRC105) to CD105
Drug: Sorafenib — 400 mg of sorafenib will be given twice daily.
  Other Names: Nexavar

SUMMARY:
The purpose of the phase 1b portion is to evaluate safety and tolerability and determine a recommended phase 2 dose for TRC105 when added to standard dose sorafenib in patients with hepatocellular carcinoma. Up to 18 patients will be treated.

The purpose of the phase 2 portion is to estimate the ORR of patients with hepatocellular carcinoma by RECIST 1.1. Up to 21 patients will be treated in phase 2.

DETAILED DESCRIPTION:
Sorafenib is an oral multikinase inhibitor targeting several receptor tyrosine kinases, including the VEGF receptor (VEGFR), implicated in pathologic angiogenesis, tumor growth, and cancer progression. Sorafenib is approved for the treatment of unresectable hepatocellular carcinoma (HCC). TRC105 is an antibody to endoglin, an important angiogenic target on proliferating endothelial cells that is distinct from VEGFR. TRC105 inhibits angiogenesis, tumor growth and metastases and complements the activity of bevacizumab and multi-kinase inhibitors that target the VEGFR in preclinical models. Together, the use of TRC105 with sorafenib may result in more effective angiogenesis inhibition and improved clinical efficacy over that seen with sorafenib alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have confirmed hepatocellular carcinoma (HCC) by histopathology or imaging criteria according to AASLD guidelines.
2. Patients must have disease that is not amenable to potentially curative resection or ablative techniques or that has recurred following ablative techniques. In addition, disease must not be amenable to transhepatic arterial chemoembolization (TACE) or must have progressed on TACE. Patients must not be candidates for liver transplantation.
3. If liver cirrhosis is present, patient must have a Child-Pugh A or B (7 points) classification.
4. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission per investigators' clinical judgment.
5. Measurable disease by RECIST 1.1 (Phase 2 only)
6. Age of 18 years or older
7. ECOG performance status ≤ 1
8. Resolution of all acute adverse events resulting from prior cancer therapies to NCI CTCAE grade ≤ 1 or baseline
9. Adequate organ function
10. Willingness and ability to consent to participate in study
11. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
12. Men who are sterile OR agree to use at least two forms of a reliable and highly effective method of birth control and to not donate sperm and for at least 180 days following last dose of TRC105 or sorafenib.
13. Woman of non-child bearing potential due to surgical sterilization confirmed by medical history or menopause, OR woman of child bearing potential who test negative for pregnancy at time of enrollment based on serum pregnancy test and agree to use at least 2 forms of a reliable and highly effective method of birth control during the study and for at least 180 days after stopping TRC105 or sorafenib.

Exclusion Criteria:

1. Prior anticancer systemic therapy
2. Current treatment on another therapeutic clinical trial
3. Prior radiation therapy within 28 days of starting the study treatment
4. No major surgical procedure or significant traumatic injury within 6 weeks prior to study registration, and must have fully recovered from any such procedure.
5. Proteinuria
6. Uncontrolled chronic hypertension defined as systolic > 150 or diastolic > 90 despite optimal therapy.
7. History of brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.
8. Angina, MI, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, PTCA or CABG within the past 6 months.
9. Active bleeding or pathologic condition that carries a high risk of bleeding. No bleeding diathesis.
10. Thrombolytic use within 10 days prior to first day of study therapy
11. History of hemorrhage or hemoptysis (> ½ teaspoon bright red blood) within 3 months of starting study treatment
12. Need for anticoagulation
13. History of liver transplant
14. History of bleeding esophageal varices in previous 6 months, which have not been adequately managed with banding or sclerotherapy.
15. History of peptic ulcer disease within 3 months of treatment.
16. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
17. Patients may not have received a strong CYP3A4 inducer within 12 days prior to registration
18. Patients with known hypersensitivity to Chinese hamster ovary products or other recombinant human, chimeric, or humanized antibodies.
19. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality
20. Ascites or pleural effusion requiring intervention or that required intervention within the last month and has recurred
21. Pericardial effusion (except trace effusion identified by echocardiogram)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Theuer, MD, PhD, Study Director — Tracon Pharmaceuticals Inc.
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - University Hospitals, Cleveland, Ohio
  - MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Carotuximab (10 mg/kg wk to 15 mg/kg Bi-wk) Plus Sorafenib: Carotuximab (TRC105) given weekly (10 mg/kg) for 2 cycles then bi-weekly iv TRC105 (15 mg/kg) with 400mg sorafenib twice daily
- Carotuximab (10 mg/kg Weekly) Plus Sorafenib: Carotuximab (TRC105) given weekly iv (10 mg/kg) with 400mg sorafenib twice daily
Period: Overall Study
Arm/Group | Carotuximab (10 mg/kg wk to 15 mg/kg Bi-wk) Plus Sorafenib | Carotuximab (10 mg/kg Weekly) Plus Sorafenib
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients who received at least a portion of a dose of Carotuximab
Groups:
- Total: Total of all reporting groups
Arm/Group | Carotuximab (10 mg/kg wk to 15 mg/kg Bi-wk) Plus Sorafenib | Carotuximab (10 mg/kg Weekly) Plus Sorafenib | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 14 | 9 | 23
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2 | 0 | 2
  White | 9 | 7 | 16
  Black or African American | 2 | 5 | 7
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experience Dose Limiting Toxicities by Dose Level
Description: If 1 of 3 patients experienced a DLT, the dose level was expanded to 6 patients. The maximum tolerated dose (MTD) would have been exceeded if ≥ 33% of patients experience DLT at a given dose level. DLT occurred when a patient had 1 or more toxicities outlined in the protocol that was considered at least possibly related to TRC105 during the first 4 months of participation in the trial. The number of DLTs by dose cohort have been presented.
Time Frame: 4 months
Population: Patients must have received at least a portion of a dose of TRC105 or sorafenib to be evaluable for assessment of DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Carotuximab (10 mg/kg wk to 15 mg/kg Bi-wk) Plus Sorafenib | Carotuximab (10 mg/kg Weekly) Plus Sorafenib
Number analyzed (Participants) | 14 | 13
Participants | 1 | 0

2. Primary Outcome: Overall Response Rate (ORR)
Description: Number of patients with a response (PR or CR) are included by dose level. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Patients must have had a screening scan and at least 1 on study scan to be eligible for RECIST 1.1 evaluation.
Time Frame: 4 months
Population: Patients must have had a screening scan and at least 1 on study scan to be eligible for RECIST 1.1 evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Carotuximab (10 mg/kg wk to 15 mg/kg Bi-wk) Plus Sorafenib | Carotuximab (10 mg/kg Weekly) Plus Sorafenib
Number analyzed (Participants) | 14 | 11
Participants | 2 | 1

3. Secondary Outcome: Pharmacokinetic Profile of TRC105 When Given With Sorafenib
Description: Steady state mean trough serum concentrations by dose level of TRC105 after 5 weeks of dosing were measured using validated methods after 5 weeks of dosing.
Time Frame: 5 weeks
Population: Steady state mean trough serum concentration by dose level after 5 weeks of dosing. Patients must have received all protocol required TRC105 doses to be included in the analysis. Additional analysis were not performed as TRC105 development overall was canceled due to lack of efficacy.
Measure: Mean (Standard Deviation); unit: ug/ML
Arm/Group | Carotuximab (10 mg/kg wk to 15 mg/kg Bi-wk) Plus Sorafenib | Carotuximab (10 mg/kg Weekly) Plus Sorafenib
Number analyzed (Participants) | 8 | 3
ug/ML | 14.2 (12.1) | 44.7 (9)

4. Secondary Outcome: TRC105 Immunogenicity as Assessed by Anti-Product Antibody (APA)
Description: Number of patients who tested positive for antibodies to TRC105 by dose level. Anti-Product Antibody (APA) concentrations were measured using validated ELISA methods.
Time Frame: 19 months
Population: Number of patients who tested positive for antibodies to TRC105. Patients must have tested negative for TRC105 antibodies at baseline and have had an on study test performed to be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Carotuximab (10 mg/kg wk to 15 mg/kg Bi-wk) Plus Sorafenib | Carotuximab (10 mg/kg Weekly) Plus Sorafenib
Number analyzed (Participants) | 13 | 5
Participants | 9 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected while on study and for 28 days following the last dose of TRC105 or sorafenib. The longest duration of participation of any patient on study was 24 months.
Description: Only patients who received at least a portion of a dose of TRC105 or sorafenib were included in the safety population. Both dose groups received 10 mg/kg TRC105 for the first month. Patients assigned to the 10 mg/kg weekly (cycle 1) then 15 mg/kg every two weeks (cycle 2+) dose group who discontinued the study prior to initiating cycle 2 dosing were counted in the 10 mg/kg weekly adverse event group.
Arm/Group | Carotuximab (10 mg/kg wk to 15 mg/kg Bi-wk) Plus Sorafenib | Carotuximab (10 mg/kg Weekly) Plus Sorafenib
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 5/14 | 9/13
Other Adverse Events (participants affected / at risk) | 14/14 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carotuximab (10 mg/kg wk to 15 mg/kg Bi-wk) Plus Sorafenib (N=14) | Carotuximab (10 mg/kg Weekly) Plus Sorafenib (N=13)
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Aspartate Aminotransferase Increase (Investigations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Epstaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Oesophageal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Wound Infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carotuximab (10 mg/kg wk to 15 mg/kg Bi-wk) Plus Sorafenib (N=14) | Carotuximab (10 mg/kg Weekly) Plus Sorafenib (N=13)
Abdominal Pain (Gastrointestinal disorders) | 1 | 5
Abdominal Distension (Gastrointestinal disorders) | 0 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2
Agitation (Psychiatric disorders) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 3 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Ammonia Increased (Investigations) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 6 | 6
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bacteraemia (Infections and infestations) | 1 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 4
Blood Amylase Increased (Investigations) | 4 | 3
Blood Bilirubin Increased (Investigations) | 2 | 4
Blood Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 2
Blood Phosphorus Decreased (Investigations) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Chest Pain (General disorders) | 1 | 1
Chills (General disorders) | 4 | 7
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 4 | 6
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Depression (Psychiatric disorders) | 3 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 9
Dizziness (Nervous system disorders) | 1 | 3
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Eye Pain (Eye disorders) | 1 | 0
Faeces Discoloured (Gastrointestinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 3
Fatigue (General disorders) | 7 | 13
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 1
Gait Disturbance (General disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 3
Gingival Bleeding (Gastrointestinal disorders) | 2 | 5
Glossodynia (Gastrointestinal disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 11
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypertension (Vascular disorders) | 4 | 8
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Hypotension (Vascular disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 2 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 4 | 4
Insomnia (Psychiatric disorders) | 2 | 2
International Normalised Ratio Increased (Investigations) | 0 | 1
Irritability (General disorders) | 1 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Lactic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Lip Swelling (Gastrointestinal disorders) | 1 | 0
Lipase Increased (Investigations) | 4 | 4
Lung Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malaise (General disorders) | 0 | 1
Medical Device Site Bruise (General disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Microcytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 2
Mucosal Inflammation (General disorders) | 2 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 5
Neuropathy Peripheral (Nervous system disorders) | 1 | 1
Neutrophil Count Decreased (Investigations) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oedema Peripheral (General disorders) | 2 | 3
Oropharyngeal Blistering (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 6 | 8
Paraesthesia (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1
Periodontal Disease (Gastrointestinal disorders) | 2 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1
Photopsia (Eye disorders) | 1 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Rectal Ulcer (Gastrointestinal disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Scrotal Infection (Infections and infestations) | 1 | 0
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus Tachycardia (Cardiac disorders) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Skin Abrasion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Papilloma (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 2
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Testicular Swelling (Reproductive system and breast disorders) | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Tooth Abscess (Infections and infestations) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Upper Respiratory Infection (Infections and infestations) | 1 | 1
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary Hesitation (Renal and urinary disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Viith Nerve Paralysis (Nervous system disorders) | 0 | 1
Vision Blurred (Eye disorders) | 0 | 2
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Weight Decreased (Investigations) | 2 | 3
Weight Increased (Investigations) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 1

LIMITATIONS AND CAVEATS:
TRC105 development has been discontinued due to lack of efficacy. Secondary endpoints including PFS, OS, duration of response, sorafenib PK, circulating angiogenic biomarkers and assessment of IGF-1-modified Child-Pugh score were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT02560779/Prot_SAP_000.pdf